CLINICAL TRIAL: NCT02926274
Title: Transfusion of Stored Whole Blood in a Civilian Trauma Center: A Prospective Evaluation of Feasibility and Outcomes
Brief Title: Transfusion Using Stored Whole Blood
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: NTI-JWMRP-201501
Record Dates: First submitted 2016-08-29; First posted 2016-10-06 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Trauma; Hemorrhage; Coagulopathy
Keywords: whole blood; trauma; transfusion; coagulopathy
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Whole Blood: Adult male trauma patients presenting with systolic blood pressure <100 will receive up to 6 units of whole blood when available.
- Component therapy: Adult female patients presenting with systolic blood pressure <100, as well as adult male patients with systolic blood pressure <100 during periods when whole blood is not available, will receive component therapy (1:1:1 packed red blood cells: plasma:platelets) for transfusion.

SUMMARY:
Massive hemorrhage is a major cause of potentially preventable death following trauma. A common consequence of hemorrhagic shock is uncontrollable bleeding from coagulopathy, leading to death from exsanguination. Even when bleeding is controlled, patients are at increased risk of complications and mortality. Reconstituted whole blood, or component therapy with packed red blood cells (PRBCs), plasma, and platelets was introduced by the military in recent conflicts in Iraq and Afghanistan with remarkable results and has been adopted by most civilian trauma centers. Despite improving coagulopathy, it is apparent that transfusion of blood components is not equivalent to whole blood transfusion. Transfusion of high plasma volumes may be associated with increased risk of allergic reaction, transfusion associated acute lung injury (TRALI), hypervolemic cardiac failure, and acute respiratory distress syndrome (ARDS). Military services have recently reintroduced fresh whole blood (WB) for standard resuscitation of massive hemorrhage, have found that WB offers a survival advantage over component therapy, and that risks of transfusion reactions are similar for WB and PRBCs. On the civilian side, whole blood is an FDA-licensed product that has been in use in pediatric open heart surgery and autologous blood donation but is no longer commonly available for other indications. However, the military results are renewing interest in whole blood for trauma resuscitation. The use of low-antibody titer whole blood leukoreduced with a platelet-sparing filter was recently approved by the University of California Los Angeles Blood and Blood Derivatives Committee and two other trauma centers for male trauma patients. This study will test the feasibility of providing stored WB for resuscitation of patients in hemorrhagic shock and determine the effects of WB on clinical outcomes as well as the effects on coagulation, fibrinolysis, and inflammation, compared to standard blood component therapy.

DETAILED DESCRIPTION:
Most current massive transfusion protocols attempt to treat the early coagulopathic state induced by severe injury and hemorrhagic shock with transfusion of red blood cells, plasma, and platelets in a 1:1:1 ratio replicating whole blood. Civilian trauma centers have now begun to initiate resuscitation of adult male patients with stored whole blood as a standard of care, however.

The main hypothesis behind this change in practice is that transfusion of whole blood (WB) rather than attempted reconstitution from its banked components is safer, more efficient and effective treatment of hemorrhagic shock following injury and will result in less frequent development of clinical coagulopathy and subsequent mortality. Whole blood offers the advantages of more precisely approximating shed blood; decreased volume of additives per unit; and exposure to a decreased number of donors for a patient undergoing massive transfusion. It remains to be seen whether this will translate into differences in coagulopathy, inflammation, and mortality. The purpose of this study is to investigate the feasibility of developing a system to collect, store, and deliver whole blood for trauma resuscitations in a civilian trauma center.

The universal donor blood type for patients with unknown blood type is type O positive blood for males and O negative for females. Because O negative blood is rare the study will initiate the change in practice in adult male patients and later extend it to female patients if feasible. The study will determine the effects of WB transfusion in adult male patients compared to transfusion of PRBCS, plasma, and platelets in a 1:1:1 ratio in non adult male patients on markers of coagulation, fibrinolysis, and inflammation, as well as the development of complications and hospital mortality following severe injury.

Specific aims are to:

1. Determine the appropriate shelf life of WB that has been leukoreduced with a platelet sparing filter by measuring changes in levels of coagulation factors and global clotting potential of banked units over time. To accomplish this the investigators will measure variables known to reflect potential and actual clotting capacity including platelet function and overall clotting ability by thromboelastography (TEG) and thrombin generation analysis in whole blood up to 35 days.
2. Prospectively determine the effectiveness of trauma resuscitation using WB compared to component therapy and its effects on variables known to reflect potential and actual clotting capacity including markers of coagulation, fibrinolysis, inflammation, platelet function and global hemostatic potential post transfusion, as well as hospital outcomes including development of coagulopathy, infection, venous thromboembolism (VTE), multiple organ failure (MOF), total transfusion requirements, and mortality.
3. Test the feasibility and implementation of a system to provide WB for resuscitation of trauma patients in hemorrhagic shock in civilian trauma centers. This will be accomplished by monitoring cost, storage needs, frequency of blood collection, number of donors, inventory, utilization and wastage of unused units.

ELIGIBILITY:
Inclusion Criteria:

* All adult trauma patients presenting to Ronald Reagan University of California Los Angeles (UCLA) Medical Center with systolic blood pressure <100 suspected due to hemorrhage are eligible. Adult males will receive whole blood when available. Adult female patients will receive component therapy.

Exclusion Criteria:

* Burn patients, patients with medical bracelets or other directives refusing blood transfusion if known during emergent resuscitation for traumatic injury, pediatric patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients presenting to Ronald Reagan UCLA Medical Center with systolic blood pressure <100 suspected due to hemorrhage are eligible. Adult males will receive whole blood when available. Adult female patients will receive component therapy.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Volume of blood products transfused during resuscitation | From admission to 24 hours after admission
  Volume of blood products transfused (whole blood, packed red blood cells, platelets, and plasma) within the first 24 hours of admission.

SECONDARY OUTCOMES:
mortality | Mortality at 30 days after injury
platelet mapping by thromboelastography | within one day of injury, after 6 units of whole blood or packed red blood cell transfusion, or after hemostasis is achieved if less than 6 units are required
  Platelet mapping determines the degree of inhibition of platelet function, measured on blood samples from patients being resuscitated during hemorrhagic shock. The primary outcome is the sample taken immediately following transfusion of 6 units of whole blood or packed red blood cells during initial resuscitation (almost always within one day of injury); or, if less than 6 units are transfused before hemostasis is achieved, immediately after transfusion of the last unit (within one day after injury).
Thromboelastography reaction time | within one day of injury, after 6 units of whole blood or packed red blood cell transfusion, or after hemostasis is achieved if less than 6 units are required
  Determines the time to first evidence of clot formation, measured on blood samples from patients being resuscitated during hemorrhagic shock. The primary outcome is the sample taken immediately following transfusion of 6 units of whole blood or packed red blood cells during initial resuscitation (almost always within one day of injury); or, if less than 6 units are transfused before hemostasis is achieved, immediately after transfusion of the last unit (within one day after injury).
Thromboelastography K value | within one day of injury, after 6 units of whole blood or packed red blood cell transfusion, or after hemostasis is achieved if less than 6 units are required
  Determines the time from first evidence of clot formation to the time the clot reaches a diameter of 20mm, thus representing the rate of clot formation. This will be measured on blood samples from patients being resuscitated during hemorrhagic shock. The primary outcome is the sample taken immediately following transfusion of 6 units of whole blood or packed red blood cells during initial resuscitation (almost always within one day of injury); or, if less than 6 units are transfused before hemostasis is achieved, immediately after transfusion of the last unit (within one day after injury).
Thromboelastography maximum amplitude (MA) | within one day of injury, after 6 units of whole blood or packed red blood cell transfusion, or after hemostasis is achieved if less than 6 units are required
  Maximum amplitude is a measure of overall clot strength measured on blood samples from patients being resuscitated during hemorrhagic shock. The primary outcome is the sample taken immediately following transfusion of 6 units of whole blood or packed red blood cells during initial resuscitation (almost always within one day of injury); or, if less than 6 units are transfused before hemostasis is achieved, immediately after transfusion of the last unit (within one day after injury).
total units of blood products transfused (includes whole blood, packed red blood cells, plasma, platelets, and cryoprecipitate). | 3 and 6 hours after admission, 24 hours after admission, and total for hospital stay within 30 days of injury
venous thromboembolism | any venous thromboembolism occurring during hospitalization within 30 days of injury.
infection (documentation of suspected or confirmed infection in the medical chart including urinary tract infection, pneumonia, wound infection, infectious colitis, and bacteremia). | during hospitalization within 30 days of injury.
Development of clinical coagulopathy | Within 24 hours of injury, and during hospitalization within 30 days
  Documentation of diffuse clinical bleeding or documented clinical coagulopathy based on laboratory evidence by the primary team
Development of Acute Respiratory Distress Syndrome | During hospitalization within 30 days
Development of acute kidney injury requiring renal replacement therapy | During hospitalization within 30 days
Hemolysis | within 24 hours of admission
  7. Hemolysis as measured by haptoglobin, bilirubin, lactate dehydrogenase, and direct antiglobulin
cerebrovascular accident | During hospitalization within 30 days
acute coronary syndrome | During hospitalization within 30 days
transfusion-related lung injury | During hospitalization within 30 days
transfusion-associated cardiac overload | During hospitalization within 30 days
Duration of need for renal replacement therapy | During hospitalization within 30 days
Duration of need for mechanical ventilation | During hospitalization within 30 days
Duration ICU admission | During hospitalization
Duration hospital admission | During hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Fully deidentified data will be available to other researchers upon request

REFERENCES:
- [Derived] Siletz AE, Blair KJ, Cooper RJ, Nguyen NC, Lewis SJ, Fang A, Ward DC, Jackson NJ, Rodriguez T, Grotts J, Hwang J, Ziman A, Cryer HM. A pilot study of stored low titer group O whole blood + component therapy versus component therapy only for civilian trauma patients. J Trauma Acute Care Surg. 2021 Oct 1;91(4):655-662. doi: 10.1097/TA.0000000000003334. PMID 34225348

DOCUMENTS (1):
  • Study Protocol (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT02926274/Prot_000.pdf